CLINICAL TRIAL: NCT07153809
Title: Randomized, Double-blind Clinical Trial on the Efficacy and Safety of Gut Microbiota Transplantation (FMT) in the Treatment of Moderate to Severe Acute Pancreatitis
Brief Title: Fecal Microbiota Transplantation (FMT) in Patients With Moderate to Severe Acute Pancreatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xiangyu Kong, Principle Investigator, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHEC2024-297
Record Dates: First submitted 2024-09-07; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Acute Pancreatitis; Severe Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Physiological saline placebo will be injected through a nasojejunal nutrition tube once a day for five days.
  Interventions: Procedure: Placebo
- FMT (Experimental): FMT bacterial solution will be injected through a nasojejunal nutrition tube once a day for five days.
  After intestinal preparation (via nasal feeding of inulin or oligofructose 24 hours before FMT), the subjects underwent 5-6 consecutive FMT treatments (injecting 100ml of standard bacterial solution 1/d into the nasojejunal nutrition tube, with a minimum of 2.5 * 1012 CFU of viable cells per 50mL of bacterial solution).
  FMT intervention can be performed when the subject's intestinal function is restored and SIRS indicators are significantly relieved compared to before.
  During the research period, long-term use of probiotics, antibiotics, and other foods and drugs that interfere with and damage gut microbiota is prohibited. Subjects need to be informed in advance before taking any medication.
  All subjects need to complete relevant examinations before enrollment. Conduct a comprehensive safety and efficacy evaluation during treatment, after treatment, and one week after treatment.
  Interventions: Procedure: FMT

INTERVENTIONS:
Procedure: FMT — FMT bacterial solution will be injected through a nasojejunal nutrition tube once a day for five days.
  Arms: FMT
Procedure: Placebo — Physiological saline placebo will be injected through a nasojejunal nutrition tube once a day for five days.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind and placebo-controlled study. The purpose of this study is to evaluate the efficacy and safety of FMT in patients with moderate to severe acute pancreatitis.

DETAILED DESCRIPTION:
This study is a single center, randomized controlled trial. After the start of the study, 80 patients with acute moderate to severe acute pancreatitis were randomly selected according to inclusion and exclusion criteria and divided into an intervention group (n=40) and a control group (n=40) to explore the safety and efficacy of FMT in preventing late complications of acute moderate to severe acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

Age: 18-70 years old Diagnosis: Meets the diagnostic criteria for severe acute pancreatitis (SAP)

* Organ function: There may be organ failure and systemic complications that can be recovered within 48 hours
* Stage of the disease: Approximately 2 weeks after onset (non acute phase), accompanied by accumulation of pancreatic fluid volume, and significant improvement in CTSI score compared to before (grade II)
* Nutritional support: Enteral nutrition tube has been left in place Feasibility of transplantation: No absolute contraindications for gut microbiota transplantation
* Informed Consent: Voluntarily sign a written informed consent form
* Gastrointestinal status:

Abdominal pressure (bladder pressure measurement)<12mmHg ◦ Existence of spontaneous defecation/exhaust Significant improvement in abdominal distension compared to before

Exclusion Criteria:

Serious complications: combined gastrointestinal bleeding or intestinal fistula

* Special population: Pregnant or lactating women
* Informed refusal: Failure to sign informed consent form
* Basic organ dysfunction: Prior to admission, there were chronic organ dysfunction in the heart, lungs, liver, kidneys, or blood system Malignant tumor: Suffering from incurable malignant tumors
* Immune abnormalities:

Autoimmune diseases

◦ Immunosuppression status (solid organ/bone marrow transplantation history, AIDS, long-term use of immunosuppressants/hormones)

* Enteral nutrition intolerance: unable to meet 50% of calorie requirements due to severe diarrhea, fibrotic intestinal stenosis, severe gastrointestinal edema, high flow intestinal fistula, etc
* Systemic infection: meets the diagnostic criteria for systemic inflammatory response syndrome (SIRS)
* Antibiotic dependence: broad-spectrum antibiotic intervention is required for combined extraintestinal organ infections
* Immunodeficiency: Congenital or acquired immunodeficiency
* Mental illness: severe mental disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pancreatic infectious complications | through study completion, an average of 1 year
  Infectious pancreatic necrosis, sepsis, and pancreatic fistula. Infectious pancreatic necrosis: (1) Imaging suggests the formation of gas at the site of necrosis aggregation; (2) Gram staining or culture positivity of necrotic specimens obtained through percutaneous fine needle aspiration (FNAC); (3) Clinically suspected infection symptoms. However, due to the high false positive rate, routine FNAC examination is not recommended.
  Sepsis: (1) Two blood cultures (or bone marrow cultures) are positive for the same pathogen. (2) Systemic inflammatory response syndrome (SIRS) occurs.
  Pancreatic fistula: (1) History of acute necrotizing pancreatitis attacks; (2) Imaging supports the diagnosis of pancreatic fistula.
  Measurement: Yes/No (incidence rate)

SECONDARY OUTCOMES:
Change in CTSI score | through study completion, an average of 1 year
  The CT Severity Score (CTSI) of acute pancreatitis can evaluate the severity of acute pancreatitis, predict the probability of complications such as organ failure in the early stages of the disease, and assess the prognosis of patients
  Method:
  Measure CTSI scores during baseline and after FMT treatment
Changes in gut microbiome community | Up to 1 week
  The average change in bacterial species relative to baseline compared to one week after fecal microbiota transplantation (FMT).
Gastrointestinal mucosal barrier index | Up to 1 weeks
  Diamine oxidase (DAO): It is a marker enzyme of intestinal mucosal cells. D-Lactic acid: It is a metabolic product of intestinal bacteria. Under normal circumstances, the content in plasma is extremely low. When the intestinal mucosa is damaged, DAO and D-lactate will be released into the blood in large quantities, leading to a significant increase in blood concentration, which is an important indicator for evaluating the structural integrity of the intestinal mucosa. During the treatment process, changes in DAO and D-lactate levels can reflect the progress of intestinal mucosal repair.
  DAO decline rate Formula: (Baseline Value -7-Day Value)/Baseline Value x 100% Unit:% D-lactic acid decline rate Formula: (Baseline Value -7-Day Value)/Baseline Value x 100% Unit:%
Markers of inflammatory conditions | Up to 3 months
  C-reactive protein (CRP) is a measure of inflammatory status and is considered a biomarker of inflammation in patients with pancreatitis.
Inflammatory markers | Up to 3 months
  Procalcitonin (PCT) is a measure of inflammatory status and is considered a biomarker of inflammation in patients with pancreatitis
Inflammatory markers | Up to 3 months
  Interleukin-6 (IL-6) is a measure of inflammatory status and is considered a biomarker of inflammation in patients with pancreatitis
Inflammatory markers | Up to 3 months
  lactic acid is a measure of inflammatory status and is considered a biomarker of inflammation in patients with pancreatitis

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China